CLINICAL TRIAL: NCT03136302
Title: Correlation of Tractography and Motor Evoked Potentials in Deep Brain Stimulation
Status: Recruiting | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: DBS2017
Record Dates: First submitted 2017-01-25; First posted 2017-05-02 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Improving Accuracy of Implanting Stimulation Electrodes
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subthalamic Nucleus (STN): Patients with Parkinson's disease
  Interventions: Procedure: Deep Brain Stimulation
- Globus Pallidus (Gpi): Patients with Dystonia
  Interventions: Procedure: Deep Brain Stimulation
- Ventral intermediate nucleus of the thalamus (VIM): Patients with Tremor
  Interventions: Procedure: Deep Brain Stimulation

INTERVENTIONS:
Procedure: Deep Brain Stimulation — Deep Brain Stimulation

SUMMARY:
The goal is to establish another anatomical referencing system in order to achieve an even higher accuracy when implanting stimulation electrodes.

DETAILED DESCRIPTION:
The main goal is to find out what are the optimal distances to these reference fiber tracts when stimulating and to find the optimal target. This has to be evaluated for each target, such as globus pallidus (Gpi), subthalamic nucleus (STN) and ventral intermediate nucleus of the thalamus (VIM) separately. This is of special importance as the investigators can demonstrate the internal capsule, which is often a generator of stimulation-induced side effects: tetanic muscle contractions, dysarthria and gaze deviations.

ELIGIBILITY:
Inclusion Criteria:

* Patient qualifying for deep brain stimulation on the basis of a movement disorder (Parkinson's Disease, tremor, dystonia) or chronic pain disease.
* Informed consent

Exclusion Criteria:

* Lack of consent
* Electrical or other devices that preclude the performance of an MRI

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who qualify for deep brain stimulation on the basis of a movement disorder and chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
distance between stimulation electrode and motor fibers in mm | Intraoperative
  Distances between the stimulation electrode and motor fibers as depicted on fiber tracking in millimeters in correlation to the threshold current for eliciting clinical side effects

SECONDARY OUTCOMES:
Intraoperative intensity of stimulation in milliampere (mA) | Intraoperative
  Intraoperative intensity of stimulation in milliamp, which elicits an activation of contralateral muscle groups (musculus interosseus dorsalis and the musculus tibialis anterior)
Stimulation thresholds in milliampere (mA) | Intraoperative
  Threshold of intraoperative stimulation intensity in milliamp, which elicits capsular side effects
Change in disease score units on the UPDRS rating scale | twelve months
  Assessment of therapeutic effects using Unified Parkinson disease rating scale (UPDRS)
Change in disease score units on the FTRS rating scale | twelve months
  Assessment of therapeutic effects using, Fahn-Tremor Rating Scale (FTRS)
Change in disease score units on the BFMDRS rating scale | twelve months
  Assessment of therapeutic effects using Burke-Fahn-Marsden dystonia rating scale (BFMDRS)
Change in disease score units on the TWSTR rating scale | twelve months
  Assessment of therapeutic effects using Toronto Western Spasmodic torticollis rating scale (TWSTR)
Change in disease score units on the PDQ-39 rating scale | twelve months
  Assessment of therapeutic effects using Parkinsons Disease QuestionnairePDQ-39

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Weise, MD, Principal Investigator — Dalhousie University
Locations (1):
- Queen Elizabeth Health Science Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided